CLINICAL TRIAL: NCT01463969
Title: High Plasma Level of Long Pentraxin 3 is Associated With Insulin Resistance in Women With Polycystic Ovary Syndrome
Brief Title: High Plasma Level of Long Pentraxin 3 is Associated With Insulin Resistance in Women With Polycystic Ovary Syndrome (PCOS)
Status: Completed | Type: Observational
Sponsor: Gulhane School of Medicine (Other)
Responsible Party: Principal Investigator, Aydogan Aydogdu, MD, Gulhane School of Medicine
Other Study IDs: 23.10.2011; 24.05.2011 (Registry Identifier: pcos and PTX3)
Record Dates: First submitted 2011-10-23; First posted 2011-11-02 (Estimated); Last update posted 2011-11-02 (Estimated); Status verified 2011-10

CONDITIONS: PCOS
Keywords: PCOS and PTX3 levels
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- PCOS patients
- Control group

SUMMARY:
In the present study, serum pentraxin 3 level and its relationship with insulin resistance were determined in patients with Polycystic Ovary Syndrome (PCOS. It was found that PTX3 level is increased in patients with PCOS and it is positively correlated with HOMA-IR.

ELIGIBILITY:
Inclusion Criteria:

* Absence of significant abnormalities on physical examination except hirsutism
* No lipid lowering, hypoglycemic, antihypertensive or hormone replacement therapy
* Normal thyroid function and prolactin level
* Absence of history or evidence of metabolic, cardiovascular, respiratory or hepatic disease

Exclusion Criteria:

* Pregnant
* Possible ovarian tumors,
* Congenital adrenal hyperplasia or
* BMI greater than 35 kg/m2

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 40 PCOS patients and 40 healty controls
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2010-05; Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Level of of pentraxin3 in cases with Polycystic Ovarian Syndrome | 1 year
  Mean PTX3 was significantly higher in patients with PCOS. This means that there is increased level of inflamation in patients with PCOS.

SECONDARY OUTCOMES:
Relationship of PTX3 with insuline resistance in patients with PCOS. | 1 year
  PTX3 was positively correlated with HOMA-IR. This means that inflamation may cause insuline resistance in patients with PCOS.

CONTACTS AND LOCATIONS:
Overall Officials: Aydogan Aydogdu, MD, Principal Investigator — Gulhane School of Medicine Dep. of Endocrinology and Metabolism
Locations (3):
- Turkey (Türkiye) (3):
  - Gulhane School of Medicine Dep. of Endocrine and Metabolism, Ankara
  - Gulhane School of Medicine Dep. of Endocrinology and Metabolism, Ankara
  - Gulhane School of Medicine, Ankara